CLINICAL TRIAL: NCT05378243
Title: Innovative Robotic Gait Trainer Use to Enable Walking in Children With Cerebral Palsy GMFCS III and IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Ontario Brain Institute (Other); Academic Health Science Centres (Other)
Responsible Party: Principal Investigator, Anna McCormick, Pediatrician / Physical Medicine and Rehabilitation Specialist, Division Chief Developmental Medicine and Rehabilitation, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20200502
Record Dates: First submitted 2022-05-05; First posted 2022-05-18 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Gait Training (Experimental): 8 weeks of therapy with the robotic gait training device 4-5 times a week for 1 hour each session
  Interventions: Device: Robotic Gait Training
- Functional Clinical Therapy (Experimental): 8 weeks of therapy with a custom designed therapy program for the participant's needs 4-5 times a week for 1 hour each session
  Interventions: Behavioral: Functional Clinical Therapy

INTERVENTIONS:
Device: Robotic Gait Training — Use of a walker adapted with robotic components to promote proper walking gait
  Arms: Robotic Gait Training
Behavioral: Functional Clinical Therapy — Personalized program of physical therapy targeted to improving walking gait
  Arms: Functional Clinical Therapy

SUMMARY:
Exploration to optimize mixed quantitative and qualitative methodology using multiple outcome measures in a randomized, cross-over trial structure comparing the effect of robotic gait training (RGT) group, and functional clinical therapy (FCT) using each subject as their own control.

DETAILED DESCRIPTION:
Exploration to optimize mixed quantitative and qualitative methodology using multiple outcome measures in a randomized, cross-over trial structure comparing the effect of robotic gait training (RGT) group, and functional clinical therapy (FCT) using each subject as their own control.

The primary objective is to assess feasibility of the study design and device tolerability. Specifically:

* Recruitment success (number screened, number eligible, number enrolled) where 80% of the recruitment target is reached.
* Attrition rates of less than 10% (i.e. ≥90% of participant's successfully complete assessments).
* Adherence for each participant: 80% of participants who complete assessments achieve the minimum target dose (i.e. approx. ≥30 hours of therapy in both study groups).
* Qualitative feedback from clinicians and patients/caregivers on device tolerability and study participation.

Secondary objectives will evaluate the distance a child can walk in two minutes using the Two Minute Walk Test (2MWT, 18) and will examine a more global impact of the use of this technology. Data collected will include quality of gait, child or proxy chosen individualized goals, hypertonicity, contractures, and bone health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cerebral palsy
* GMFCS Levels III and IV
* Ages ≥2 to ≤12 years
* Ability to take steps with and/or without assistance
* Meet the Trexo Plus device size requirements
* Ability to follow instructions and signal pain, fear, or discomfort
* Ability to safely use the device at home as determined by the study team

Exclusion Criteria:

* Lower limb or orthopedic surgery within 9 months prior to enrollment
* Botulinum toxin injections within 4 months prior to enrollment
* Serial casting within 3 months prior to enrollment
* Knee flexion contracture > 20°
* Knee valgus > 40°
* Hip subluxation > 40 % migration percentage
* Uncontrolled movements that prevent transfer in and/or out of device
* Weight bearing restrictions
* Uncontrolled seizures
* Skin lesions in areas where the device straps would be attached
* Significant language barrier with parents and/or caregivers Note: children with severe contractures will be unable to fit in the device and are therefore excluded from the study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment and recruitment in this study design | 4 months
  Recruitment success as defined by meeting 80% of the recruitment target
Retention in this study design | 4 months
  Attrition of less than 10% where 90% of participants are completing the assessments to the end of the trial
Adherance to protocol for each participant | 4 months
  Participant self-reported session diaries will be assessed to determine whether participants are achieving the min target dose of 30h of therapy over each 8 week session
Device tolerability | 4 months
  Participant caregivers will be interviewed for qualitative feedback on device/therapy tolerability after each 8 week session

SECONDARY OUTCOMES:
2 minute walk test (2mwt) | 4 months
  distance child is able to walk in their own walker in 2 minutes
Edinburgh Visual Gait Score | 4 months
  Edinburgh Visual Gait Score is used for assessing gait quality by assessing body positions and angles of various body parts through the gait pattern using a scale of 0-2 for each individual component of the assessment. A score of 0 indicates a more physiologically normal result while a score of 2 indicates a more disordered result. The scores are totaled to provide the complete score for the patient on this assessment
Physiological Cost Index | 4 months
  assessing gait efficiency by looking at the heart rate changes upon a specified exertional task. A lower physiological cost index indicates less exertion required to complete the task
Modified Ashworth Scale | 4 months
  The Modified Ashworth Scale measures resistance during passive soft tissue stretching. It is ranked by body part on a scale of 0-4 with 0 being a normal tone and 4 being highly rigid in flexion or extension.
Hypertonia Assessment Tool | 4 months
  Assessing dystonia, spasticity, and rigidity, or a mixed tone through a rating scale system where 0 indicates the behavior is not observed and 1 indicates the dystonic/spastic/rigid behavior is observed.
Barry Albright Dystonia Scale | 4 months
  Assessing dystonia and severity of dystonia in eyes, mouth, neck, trunk, each upper extremity and each lower extremity. Scored from 0-4 where 0 is an absence of dystonia and 4 is a high degree of dystonia.
Goal attainment scale | 4 months
  Attainment of self-determined goals for treatment outcomes. Goals are set with the study therapists at the outset of each treatment period and assessed using a scale of -2 to +2 where a score of 0 is the expected outcome, a negative score indicates less than expected and a positive number indicates more than expected
Spinal Alignment and Range of Motion Measure | 4 months
  Range of motion throughout the body is measured from 0-4 where 0 is no limitation and 4 is a severe limitation.
Leg Bone cortical density | 4 months
  peripheral Quantitative Computed Tomography (pQCT) Measures Cortical density (mg/cm2)
Tibia volumetric bone mineral density (BMD) | 4 months
  peripheral Quantitative Computed Tomography (pQCT) Measures Tibia volumetric bone mineral density (BMD) (mg/cm2)
Leg bone cortical cross-sectional area | 4 months
  peripheral Quantitative Computed Tomography (pQCT) Measures cortical cross-sectional area (mm2)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no intention to share IPD with other researchers